CLINICAL TRIAL: NCT00942890
Title: Strength, Pain and Function in Operation Iraqi Freedom/Operation Enduring Freedom Amputees: A Nurse-Managed Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TSNRP Grant HU0001-08-1-TS10
Record Dates: First submitted 2009-07-15; First posted 2009-07-21 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2015-10

CONDITIONS: Traumatic Amputation
Keywords: Case Management; Amputation; Muscle strength; phantom limb pain
MeSH Terms: conditions — Amputation, Traumatic; Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMES plus Standard Rehab Protocol (Experimental): NMES (EMPI 300PV stimulator) plus standard of care intervention. NMES is to the quadriceps muscle of the residual and intact limb plus rehabilitation. Therapy is 12-wks of NMES home training w/ the EMPI 300PV muscle stimulator. Participants perform training at home for 5days/wk; sessions consisted of 15 to 20 min. of NMES to each leg eliciting15 contractions/leg (10 seconds on:50 seconds off), plus a 5-minute patient treatment log, 5x/wk for 12-wks. Each contraction will be elicited by an electrical impulse generated by a battery-operated device. Two 3" X 5" electrodes are placed over the quadriceps muscle group. Participants will train at 30-40% of MVC during weeks 1-6, and 40-50% of MVC during weeks 7-12; incremental increases will be made at the study visits.
  Interventions: Device: NMES (EMPI 300PV stimulator) plus standard of care
- Standard Rehab Protocol (Active Comparator): TMARP standard of care intervention: 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1 week after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for about 6 weeks, preparing for the prosthetic. After pre-prosthetic training, patients are fitted with their prosthetic leg and began post-prosthetic training with PT. The training focus is lower limb prosthetic proficient in ambulation.
  Interventions: Behavioral: TMARP standard of care

INTERVENTIONS:
Device: NMES (EMPI 300PV stimulator) plus standard of care — In addition to the standard rehabilitation, the NMES treatment group will receive neuromuscular electrical stimulation to the quadriceps muscle of the residual and intact limb. The name of the NMES device is EMPI 300PV. NMES training will consist of performing 15 to 20 minute stimulation sessions with a 5-minute patient treatment log, 5 times per week for 12 weeks. During each training session, 15 NMES contractions per leg will be completed. Each contraction will be elicited by an electrical impulse (300PV) generated by a battery-operated device. This will be performed at home.
  Other Names: EMPI 300PV neuromuscular stimulator
  Arms: NMES plus Standard Rehab Protocol
Behavioral: TMARP standard of care — The usual care is 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1week after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for about 6 weeks, preparing for the prosthetic. After pre-prosthetic training, patients are fitted with their prosthetic leg and began post-prosthetic training with PT. The training focus is lower limb prosthetic proficient in ambulation.
  Other Names: Traditional Military Amputee Rehabilitation Program
  Arms: Standard Rehab Protocol

SUMMARY:
The purpose of this randomized control study is to determine if administering neuromuscular electrical stimulation (NMES) to the thigh muscles of a below the knee amputee is more effective than the current standard of care in preserving thigh muscle strength. In addition, this study will examine the NMES treatment effects on the participant's gait, quality of life, functional performance of standing, walking, and stair climbing, and symptoms associated with residual and phantom limb pain. The primary aim is to compare NMES plus standard rehabilitation (treatment group) to the standard rehabilitation (control group) by measuring lower extremity muscle strength. The secondary aims are to compare NMES treatment group to the control group by measuring Quality of Life (QOL) and the symptoms associated with residual & phantom limb pain. In addition to the specific aims, this study will also examine the two groups for functional performance and gait patterns after prosthetic fitting.

DETAILED DESCRIPTION:
Traumatic amputation is one of the major injuries seen as a result of Operation Iraqi and Enduring Freedom with the majority being single trans-tibial amputations (TTA). TTA experience significant reductions in thigh muscle strength of the amputated limb during the first year after amputation. The residual limb is less active in daily functions of standing and walking, resulting in progressive atrophy of the quadriceps muscles in terms of a decrease in thigh diameter which is estimated at 25% of pre-amputation diameter. An intervention that may be useful in TTA rehabilitation is neuromuscular electrical stimulation (NMES). The overall objectives of this study is to test two different approaches to prosthetic rehabilitation as potential treatments for improving muscle strength, pain and functional performance of daily activities in military personnel with TTA. Our central hypothesis is that a Nurse Managed NMES rehabilitation program will have greater improvements in muscle strength and pain as compared to the standard rehabilitation protocol alone. The rationale for this study is that NMES could have an additive effect to the Walter Reed Army Medical Center (WRAMC) standard of care program with greater improvements in muscle strength thus enhancing the performance of daily activities, Quality of Life (QOL), and decreasing disability. Such outcomes will ultimately result in decreased economic costs, accelerated rehabilitation, and potentially increase the possibility of these warriors returning to duty. The specific aims are to test Nurse Managed NMES relative to standard rehabilitation by comparing: (1) Lower extremity muscle strength; (2) QOL; and (3) Symptoms associated with phantom pain. In addition to the above aims, specific aims for the post prosthetic phase of the intervention are to compare the two groups for (4) functional performance of daily activities. After pre-testing, participants aged 18 to 55 yrs with a traumatic TTA will be randomly assigned to either the 1) Nurse Managed NMES rehabilitation program (n=30); or 2) WRAMC Amputee Protocol (n=30). Those in the NMES group will receive 12 weeks of electrical muscle stimulation 15 min/day, 5 days a week for 12 weeks. Both groups will receive the standard 12-week Walter Reed Army Medical Center rehabilitation protocol. Generalized Estimating Equation methods will be used to build regression models for statistical analysis of the longitudinal data. The significance of this research is that Nurse Managed NMES may be very important for accelerating the rehabilitation of amputees so they can achieve functional independence and regain lost muscle strength in preparation for return to duty.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral trans-tibial amputee;
2. Military service member at the time of injury (Active Duty, Reserves or National Guard);
3. Age ≥18 and ≤55 years; and
4. Able to provide freely given informed consent.

Exclusion Criteria:

1. A significant co-morbid medical condition (such as severe uncontrolled hypertension (over 160/100 mmHg) or neurological disorders such as epilepsy) where NMES strength training is contraindicated and/or participation would pose a safety threat or impair their ability to participate;
2. Unable to speak and read English;
3. Implanted cardiac pacemaker or defibrillator;
4. Vision impairment where participant is classified as legally blind (we define legally blind both clinically and functionally. Clinically, it is central visual acuity of 20/200 or less in the better eye with corrective glasses. Functionally, the participant is not able to see the digital numbers on the NMES device with corrective glasses);
5. Unwillingness to accept random assignment;
6. Currently participating in another research study with an intervention that would potentially confound the outcome variables of this study (we will also instruct participants that joining a study after being enrolled in this protocol is also not allowed); and
7. Conflicting co-morbidities including traumatic brain injury (score < 14 on glasgow coma scale), and a contralateral lower extremity injury that causes antalgic gait, pain > 5/10 consistently on the contralateral limb and/or a grade of < 4+/5 in lower extremity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Talbot, PhD, Principal Investigator — UTHSC; Michelle Kane, PhD, Principal Investigator — Walter Reed National Military Medical Center; Michael Rosenthal, PhD, Principal Investigator — Navy Medical Center San Diego
Locations (3):
- United States (3):
  - Navy Medical Center, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talbot LA, Brede E, Price M, Metter EJ. Health-related quality of life in active duty military: A secondary data analysis of two randomized controlled trials. Nurs Outlook. 2017 Sep-Oct;65(5S):S53-S60. doi: 10.1016/j.outlook.2017.07.010. Epub 2017 Jul 25. PMID 28830632
- [Derived] Talbot LA, Brede E, Metter EJ. Effects of Adding Neuromuscular Electrical Stimulation to Traditional Military Amputee Rehabilitation. Mil Med. 2017 Jan;182(1):e1528-e1535. doi: 10.7205/MILMED-D-16-00037. PMID 28051969

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a total of 44 participants.
Groups:
- Standard Rehabilitation Protocol: The usual care is 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1 wk after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for about 6 weeks, preparing for the prosthetic. After pre-prosthetic training, patients are fitted with their prosthetic leg and began post-prosthetic training with PT. The training focus is lower limb prosthetic proficient in ambulation.
- NMES Plus Standard Rehabilitation Protocol: NMES (EMPI 300PV stimulator) plus TMARP standard of care intervention. NMES is to the quadriceps muscle of the residual and intact limb plus rehabilitation. Therapy is 12-wks of NMES home training w/ the EMPI 300PV muscle stimulator. Participants perform training at home for 5days/wk; sessions consisted of 15 to 20 min. of NMES to each leg eliciting15 contractions/leg (10 seconds on:50 seconds off), plus a 5-minute patient treatment log, 5x/wk for 12-wks. Each contraction will be elicited by an electrical impulse generated by a battery-operated device. Two 3" X 5" electrodes are placed over the quadriceps muscle group. Participants will train at 30-40% of MVC during weeks 1-6, and 40-50% of MVC during weeks 7-12; incremental increases will be made at the study visits.
Period: Overall Study
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Rehabilitation Protocol: The usual care is 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1week after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for about 6 weeks. After pre-prosthetic training, patients are fitted with their prosthetic leg and began post-prosthetic training with PT. The training focus is lower limb prosthetic proficient in ambulation.
- Total: Total of all reporting groups
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.3) | 26.5 (5.9) | 26.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Muscle Strength- Extension
Description: Muscle strength was measured with a handheld dynamometer for extensor knee strength of the residual and intact limb.
Time Frame: 0, 3, 6, 9, 12 wks
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- Standard Rehabilitation Protocol: The usual care is 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1 week after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for about 6 weeks. After pre-prosthetic training, patients are fitted with their prosthetic leg and began post-prosthetic training with PT. The training focus is lower limb prosthetic proficient in ambulation.
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
Kilograms
  Residual Limb: Week 0 | 24.5 (10.7) | 26.4 (13.4)
  Residual Limb: Week 3 | 27.6 (12.5) | 34.1 (12.7)
  Residual Limb: Week 6 | 33.8 (17.3) | 36.9 (12.6)
  Residual Limb: Week 9 | 35.7 (14.0) | 39.1 (16.5)
  Residual Limb: Week 12 | 36.1 (15.4) | 42.8 (14.8)
  Intact Limb: Week 0 | 45.7 (23.8) | 45.4 (17.6)
  Intact Limb: Week 3 | 45.2 (24.3) | 41.4 (16.1)
  Intact Limb: Week 6 | 45.0 (19.5) | 45.2 (13.7)
  Intact Limb: Week 9 | 46.0 (16.7) | 45.7 (16.1)
  Intact Limb: Week 12 | 49.0 (20.7) | 51.8 (16.6)
Statistical Analysis 1: Comparison: Standard Rehabilitation Protocol vs NMES Plus Standard Rehabilitation Protocol; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 0.90, Standard Error of Mean 0.24

2. Primary Outcome: Lower Extremity Muscle Strength- Flexion
Description: Muscle strength was measured with a handheld dynamometer for extensor and flexor knee strength of the residual and intact limb.
Time Frame: 0, 3, 6, 9, 12 wks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
Kilograms
  Residual Limb: Week 0 | 14.8 (8.5) | 14.2 (6.2)
  Residual Limb: Week 3 | 14.8 (7.4) | 16.7 (7.0)
  Residual Limb: Week 6 | 16.8 (7.3) | 18.7 (6.9)
  Residual Limb: Week 9 | 18.4 (7.5) | 19.9 (7.6)
  Residual Limb: Week 12 | 19.5 (8.4) | 21.8 (6.6)
  Intact Limb: Week 0 | 25.4 (7.1) | 27.8 (10.7)
  Intact Limb: Week 3 | 27.1 (10.2) | 28.7 (9.4)
  Intact Limb: Week 6 | 26.9 (10.9) | 32.2 (10.3)
  Intact Limb: Week 9 | 28.8 (9.9) | 30.9 (9.7)
  Intact Limb: Week 12 | 28.8 (10.1) | 29.4 (9.9)

3. Primary Outcome: Lower Extremity Mobility-Distance
Description: Mobility was measured by the distance walked in 2 minutes.
Time Frame: 6, 12 wks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
inches
  Usual Pace: Week 6 | 5081 (2324) | 4452 (1949)
  Usual Pace: Week 12 | 5853 (2420) | 5657 (1919)
  Fast Pace: Week 6 | 7308 (2557) | 6369 (2316)
  Fast Pace: Week 12 | 8116 (2763) | 7692 (2072)

4. Primary Outcome: Lower Extremity Mobility- Up and Go
Description: Mobility was measured by the time to complete an "up and go" test.
Time Frame: 6, 12 wks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
Seconds
  Week 6 | 7.3 (3.9) | 7.7 (4.8)
  Week 12 | 6.3 (3.5) | 7.1 (4.4)

5. Primary Outcome: Lower Extremity Mobility- Stair Climb
Description: Mobility was measured by the time to complete a timed stair climb.
Time Frame: 6, 12 wks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
Seconds
  Week 6 | 7.8 (3.8) | 7.5 (4.4)
  Week 12 | 4.7 (3.3) | 5.6 (4.0)

6. Primary Outcome: Lower Extremity Mobility-Chair Rise
Description: Mobility was measured by the number of stands during the 30-second chair rise test.
Time Frame: 6, 12 wks
Measure: Mean (Standard Deviation); unit: Number of stands
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
Number of stands
  Week 6 | 18.1 (11.4) | 15.7 (8.4)
  Week 12 | 21.7 (9.9) | 19.4 (9.2)

7. Secondary Outcome: Pain Severity
Description: Pain severity was measured using a 4-item subscale of the Brief Pain Inventory. Pain is assessed at its "worst," "least," "average," and "current" level. Scores range from 0 (no pain) to 10 (pain, as bad as one can imagine). A mean pain score was calculated from the four items.
Time Frame: 0, 3, 6, 9, 12 wks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
units on a scale
  Week 0 | 2.9 (1.5) | 3.3 (1.6)
  Week 3 | 2.6 (1.4) | 2.4 (1.6)
  Week 6 | 2.2 (1.7) | 2.2 (1.4)
  Week 9 | 2.2 (1.6) | 2.6 (1.7)
  Week 12 | 1.8 (1.6) | 2.4 (1.9)
Statistical Analysis 1: Comparison: Standard Rehabilitation Protocol vs NMES Plus Standard Rehabilitation Protocol; Test type: Superiority or Other; p < 0.05, Regression, Linear

8. Secondary Outcome: Pain Interference
Description: Pain interference was measured as how pain hindered daily activities: general activities, walking, work, mood, enjoyment of life, relations with others, and sleep using the Brief Pain Inventory. Participants rate each item on a scale from 0-10 (0=does not interfere; 10=completely interferes). The interference score represents the mean of the seven items.
Time Frame: 0, 3, 6, 9, 12 wks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Rehabilitation Protocol | NMES Plus Standard Rehabilitation Protocol
Number analyzed (Participants) | 21 | 23
units on a scale
  Week 0 | 2.9 (2.4) | 3.1 (2.4)
  Week 3 | 2.5 (2.2) | 2.2 (2.0)
  Week 6 | 2.3 (2.6) | 2.4 (2.3)
  Week 9 | 2.0 (2.5) | 2.8 (2.7)
  Week 12 | 2.1 (2.5) | 2.7 (2.8)

ADVERSE EVENTS:
Groups:
- Standard Rehabilitation Protocol: The usual care is 12 weeks of the Traditional Military Amputee Rehabilitation Program (TMARP). TMARP training starts 1-week after surgical closure of the residual limb. Physical Therapy performs Pre-Prosthetic Training for ~6 weeks, preparing for the prosthetic. After pre-prosthetic training, patients are fitted with the prosthetic leg and began post-prosthetic training. The training focus is lower limb prosthetic proficient in ambulation.
  NMES (EMPI 300PV) plus standard of care: In addition to the standard rehabilitation, the NMES group will receive NMES to the quadriceps muscle of the residual & intact limb. The name of the NMES device is EMPI 300PV. NMES training will consist of 15-20 minute stimulation sessions with a 5-minute patient treatment log, 5 times/week for 12 weeks. During each session, 15 NMES contractions/leg will be completed. Each contraction will be elicited by an electrical impulse (300PV) generated by a battery-operated device. This will be performed at home.
- NMES w/ Rehab: The treatment group receives NMES to the quadriceps muscle of the residual & intact limb plus rehabilitation. The therapy consists of 12-weeks of NMES using the EMPI 300PV muscle stimulator. Participants train at home for 5 days/week; each session consisted of 15-20 min of NMES to each leg eliciting 15 contractions/leg (10 sec on:50 sec off), plus a 5-min tx log. Participants will train at 30-40% of MVC during weeks 1-6, and 40-50% of MVC during weeks 7-12; incremental.
  NMES plus standard of care: In addition to the standard rehabilitation, the NMES treatment group will receive NMES to the quadriceps muscle of the residual & intact limb. EMPI 300PV is the NMES device. NMES training will consist of performing 15-20 minute stimulation sessions with a 5-minute patient tx log, 5 times/week for 12 weeks. During each session, 15 NMES contractions/leg will be completed at home. Each contraction will be elicited by an electrical impulse (300PV) generated by a battery-operated device.
Arm/Group | Standard Rehabilitation Protocol | NMES w/ Rehab
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

LIMITATIONS AND CAVEATS:
The limitations of the the study was that it was not powered to detect a small or moderate difference between the two treatment groups. The sample was small and limited to military service members.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No